CLINICAL TRIAL: NCT01605448
Title: Mindfulness Based Stress Reduction for Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Rebecca Wells, Instructor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P-000411
Record Dates: First submitted 2012-05-13; First posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Alzheimer's disease; Meditation; Default Mode Network
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR (Experimental): Mindfulness Based Stress Reduction
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Control Group (No Intervention): Continue in Usual care; offered the intervention at the end of the study

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — 8 weekly classes of meditation/yoga
  Arms: MBSR

SUMMARY:
The investigators are investigating the benefits of a mind/body intervention, Mindfulness Based Stress Reduction, for adults with Mild Cognitive Impairment.

DETAILED DESCRIPTION:
We propose a prospective, randomized controlled pilot trial assessing the feasibility and safety of a study investigating mindfulness based stress reduction (MBSR) as an intervention in adults with Mild Cognitive Impairment (MCI). We are assessing safety and feasibility of this intervention, as well as using neuroimaging (fMRI) to assess improved connections in the default mode network. We will also be assessing the impact of this intervention on cognitive function and measures of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MCI* made by a neurologist (through history, physical exam and neuropsychological testing)

  1. Memory complaint, corroborated by an informant
  2. Abnormal memory function documented by memory testing <1.5 standard deviation below normative controls (assessed with the Wechsler Memory scale IV[114], Logical Memory subtest, or an equivalent test)
  3. Normal general cognitive function
  4. Mini-Mental Status Exam (MMSE) score of >24 out of 30
  5. No/minimal impairment in activities of daily living
  6. Not sufficiently impaired, cognitively or functionally, to meet the National Institute of Neurological and Communicative Disease and Stroke/Alzheimer's Disease and Related Disorders Association criteria for AD
* 60-90 yo
* Clinical Dementia Rating (CDR total score of 0.5, with at least 0.5 on memory subscale
* No history of significant cerebrovascular disease based on Modified Hachinski score ≤ 4
* Hamilton Depression Rating Scale score ≤12 (to rule out depression as a contributing cause of cognitive decline)
* Able and willing to attend weekly sessions and willing to participate in daily mindfulness assignments, up to 45 min/day
* Agreeable to participate and to be randomized to either group
* Fluent in English (since the treatment groups will be run in English)
* Adequate visual and auditory acuity to allow neuropsychological testing
* Good general health with no additional diseases expected to interfere with the study
* MRI/CT scan within 24 months without indication of infection, infarction, or focal lesions.
* Family member/close friend ("informant") able to corroborate participant's history of memory loss
* Participants may take stable doses (stable for at least 4 weeks prior to screening) of certain medications including:

  * Antidepressants (except those with significant anticholinergic side effects such as tricyclic antidepressants). Patients cannot be currently depressed and or have a history of major depression within the past 2 years
  * Cholinesterase inhibitors and memantine

Exclusion Criteria:

* Actively practicing meditation and/or yoga or have taken a meditation/yoga class in the last 6 months
* Any major systemic illness or unstable medical condition which could lead to difficulty complying with the protocol, including the diagnosis of major depression
* On psychoactive medications (antidepressants with anticholinergic effects, ie. tricyclic antidepressants, neuroleptics, chronic anxiolytics, sedative hypnotics, other anticholinergics); participants may take stable doses (stable for at least 6 months) of low doses of psychoactive medicines (i.e. ≤ 1mg klonipin/day or ≤25mg Benadryl/day)
* Psychotic features, agitation, or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol
* History of alcohol or substance abuse or dependence within the past 2 years
* Any history of brain lesions or major head trauma
* Participant unable/unwilling to follow the protocol or return for follow-up
* Investigational agents prohibited at entry and for the duration of the trial
* Participation in other clinical studies involving neuropsychological measures being collected more than one time per year
* MRI exclusions: presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 8 weeks
  Participants will inform us if they have had any adverse events during the study period and we will track to see if any occur for any of the participants
Feasibility: 85% completion | 8 weeks
  To judge the feasibility of the trial, recruitment efforts will be documented in terms of number of eligible patients approached, number who declined participation, number successfullyl recruited, and number who completed the trial. The trial will be feasible if 85% (the absolute percentage of patients) complete the trial.

SECONDARY OUTCOMES:
Change in fMRI Resting state | Change from baseline to 8 weeks
  Assessing fMRI resting state to assess if there are improved connections in the default mode network (between the posterior cingulate cortex, the medial prefrontal cortex, and the hippocampus) after participating in MBSR
Change in Cognition | Change from baseline to 8 weeks
  Assessing if there are any improvements in cognition (global functioning, episodic memory, attention, executive function, and language) after adults participate in MBSR.
Change in Measures of "well-being" | Change from baseline to 8 weeks
  Assessing if there is any improvement in measures of well-being (quality of life, stress, anxiety, depression, rumination, neuroticism, optimism, hope, resilience, and mindfulness) after participating in MBSR
Qualitative Improvements | 8 weeks
  Semi-structured interviews will be conducted to assess if any qualitative improvements

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States